CLINICAL TRIAL: NCT05599425
Title: Development of a Personalized Intervention to Motivate Health Behavior Change in Midlife Adults at Risk for Alzheimer's Disease
Brief Title: Health Behavior Change in Midlife Adults at Risk for Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21AG075328 (NIH)
Record Dates: First submitted 2022-10-19; First posted 2022-10-31 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Living Education (Active Comparator): The basic healthy living education intervention is a 24-session program (two sessions/week for 12 weeks) designed to educate participants about major modifiable risk factors for Alzheimer's disease. The first session each week is didactic, intended to increase knowledge about each Alzheimer's disease risk factor. The second session involves repetition and practice of didactic material as well as strategizing cues to action
  Interventions: Behavioral: Basic Healthy Living Education
- Enhanced Healthy Living Education (Experimental): The enhanced healthy living education intervention will include the same didactic content as the basic HLE course for the first session each week. The second session will focus on personal health beliefs and how they affect specific health behaviors. This may include discussing perceived benefits, troubleshooting barriers to action, making specific action plans, and implementing natural reward systems to bolster self-efficacy.
  Interventions: Behavioral: Enhanced Healthy Living Education

INTERVENTIONS:
Behavioral: Enhanced Healthy Living Education — 24-session healthy living education program, with enhanced content about health beliefs and mechanisms of behavior change
  Arms: Enhanced Healthy Living Education
Behavioral: Basic Healthy Living Education — 24-session healthy living education program
  Arms: Healthy Living Education

SUMMARY:
Modifying health behaviors like physical activity level, diet, stress, and mental activity level can lower risk for Alzheimer's disease, but many middle-aged and older adults find it difficult to sustain health behavior changes over the long term. This project will develop a new intervention that educates people about Alzheimer's disease risk factors and helps them understand how their personal health beliefs may prevent them from making long-lasting lifestyle changes. The goal is to help people sustain health behavior changes to prevent or delay the onset of Alzheimer's disease and related dementias.

ELIGIBILITY:
Inclusion Criteria:

* age 45-69 years
* normal cognition (Minnesota Cognitive Acuity Scale > 52)
* English language fluency
* at least two of the following: i) BMI > 24.9; ii) systolic blood pressure > 125 mmHg; iii) LDL cholesterol > 115 mg/dL; iv) HbA1C > 6.0%; v) at least one APOE ε4 allele; vi) first-degree relative with AD.

Exclusion Criteria:

* history of serious mental illness (i.e., schizophrenia, bipolar disorder)
* history of neurologic or neurodevelopmental disorder
* current alcohol or drug use disorder based on self-report
* current enrollment in an AD prevention clinical trial.

Ages: 45 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Perceived Threat of Alzheimer's Disease Scale | baseline
  7-item Likert-type scale assessing perceived likelihood, concern, and consequences of Alzheimer's disease; higher scores indicate greater perceived threat
Perceived Threat of Alzheimer's Disease Scale | 4 weeks
  7-item Likert-type scale assessing perceived likelihood, concern, and consequences of Alzheimer's disease; higher scores indicate greater perceived threat
Perceived Threat of Alzheimer's Disease Scale | 8 weeks
  7-item Likert-type scale assessing perceived likelihood, concern, and consequences of Alzheimer's disease; higher scores indicate greater perceived threat
Perceived Threat of Alzheimer's Disease Scale | 12 weeks (treatment endpoint)
  7-item Likert-type scale assessing perceived likelihood, concern, and consequences of Alzheimer's disease; higher scores indicate greater perceived threat
Dementia Awareness Questionnaire | baseline
  self-report measure of knowledge of modifiable Alzheimer's disease risk factors; higher scores are associated with greater dementia awareness
Dementia Awareness Questionnaire | 4 weeks
  self-report measure of knowledge of modifiable Alzheimer's disease risk factors; higher scores are associated with greater dementia awareness
Dementia Awareness Questionnaire | 8 weeks
  self-report measure of knowledge of modifiable Alzheimer's disease risk factors; higher scores are associated with greater dementia awareness
Dementia Awareness Questionnaire | 12 weeks
  self-report measure of knowledge of modifiable Alzheimer's disease risk factors; higher scores are associated with greater dementia awareness
Generalized Self-Efficacy Scale | baseline
  10-item self-report questionnaire assessing belief in one's own abilities; higher scores indicate greater self-efficacy
Generalized Self-Efficacy Scale | 4 weeks
  10-item self-report questionnaire assessing belief in one's own abilities; higher scores indicate greater self-efficacy
Generalized Self-Efficacy Scale | 8 weeks
  10-item self-report questionnaire assessing belief in one's own abilities; higher scores indicate greater self-efficacy
Generalized Self-Efficacy Scale | 12 weeks
  10-item self-report questionnaire assessing belief in one's own abilities; higher scores indicate greater self-efficacy

SECONDARY OUTCOMES:
Mediterranean Diet Assessment Tool | baseline
  14-item measure of adherence to a Mediterranean type diet; higher scores indicate greater diet adherence
Mediterranean Diet Assessment Tool | 12 weeks
  14-item measure of adherence to a Mediterranean type diet; higher scores indicate greater diet adherence
CHAMPS Activities Questionnaire for Older Adults | baseline
  self-report measure of engagement in physical activities, tailored to older adult population; higher scores indicate greater engagement in physical activity
CHAMPS Activities Questionnaire for Older Adults | 12 weeks
  self-report measure of engagement in physical activities, tailored to older adult population; higher scores indicate greater engagement in physical activity
Florida Cognitive Activities Scale | baseline
  25-item self-report measure about engagement in mentally stimulating activities; higher scores indicate greater cognitive activity
Florida Cognitive Activities Scale | 12 weeks
  25-item self-report measure about engagement in mentally stimulating activities; higher scores indicate greater cognitive activity
Perceived Stress Scale | baseline
  10-item measure that assesses perceived stress; higher scores indicate greater perceived stress
Perceived Stress Scale | 4 weeks
  10-item measure that assesses perceived stress; higher scores indicate greater perceived stress
Perceived Stress Scale | 8 weeks
  10-item measure that assesses perceived stress; higher scores indicate greater perceived stress
Perceived Stress Scale | 12 weeks
  10-item measure that assesses perceived stress; higher scores indicate greater perceived stress
Positive and Negative Affect Schedule | baseline
  20-item measure that assesses positive and negative emotional experiences, yielding two scores; higher scores indicate greater experience of positive or negative experiences, respectively
Positive and Negative Affect Schedule | 4 weeks
  20-item measure that assesses positive and negative emotional experiences, yielding two scores; higher scores indicate greater experience of positive or negative experiences, respectively
Positive and Negative Affect Schedule | 8 weeks
  20-item measure that assesses positive and negative emotional experiences, yielding two scores; higher scores indicate greater experience of positive or negative experiences, respectively
Positive and Negative Affect Schedule | 12 weeks
  20-item measure that assesses positive and negative emotional experiences, yielding two scores; higher scores indicate greater experience of positive or negative experiences, respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Korthauer LE, Rosen RK, Tremont G, Davis JD. Intervention Development for Tailored Education for Aging and Cognitive Health (TEACH) for Dementia Prevention in Midlife Adults: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Oct 16;13:e60395. doi: 10.2196/60395. PMID 39412840